CLINICAL TRIAL: NCT03223480
Title: EUS - Guided Balloon-occluded Gastrojejunostomy Bypass (EPASS) for Unresectable Malignant Gastric Outlet Obstruction.
Brief Title: EUS - Guided Balloon-occluded Gastrojejunostomy Bypass
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Tokyo Medical University (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE2017.277
Record Dates: First submitted 2017-07-19; First posted 2017-07-21 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Gastric Outlet Obstruction
MeSH Terms: conditions — Gastric Outlet Obstruction

STUDY DESIGN:
Intervention Model Description: All patients recruited will receive EUS-guided gastrojejunostomy using the double balloon occluder
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- EUS-guided gastrojejunostomy (Experimental): The procedures would be performed under conscious sedation or monitored anesthesia by a therapeutic gastroscope. The endoscope would be used to reach the site of obstruction. The stricture would be cannulated with a 0.025" or 0.035" guide-wire. The double balloon occluder would then be inserted on guidewire beyond the duodenal-jejunal flexure and the two balloons of the occluder would be inflated. A segment of duodenum/jejunum would then be occluded and saline would be injected. A linear echoendoscope would then be inserted into the stomach to guide insertion of the gastrojejunostomy stent.
  Interventions: Device: EUS-guided gastrojejunstomy

INTERVENTIONS:
Device: EUS-guided gastrojejunstomy — As listed in the arms description

SUMMARY:
Surgical gastrojejunostomy is the conventional treatment for palliating patients suffering from of inoperable malignant gastric outlet obstruction (GOO). Although, the procedure is associated with a high success and low re-intervention rates, there is a risk of morbidities (10% - 16%) and mortalities (7%). The placement of a pyloro-duodenal self-expandable metallic stent (DSEMS) is an alternative to surgery for the palliating these patients. As compared to surgery, the procedure is associated with shorter hospital stay, reduced morbidities and cost. However, the clinical efficacy of DSEMS is limited by several problems. In uncovered DSEMS, the long-term patency is reduced by tumor ingrowth leading to subsequent re-stenosis. In covered DSEMS, stent migration occurs at a frequency of 14 - 25% and it is a major obstacle to stent patency. As a result, randomized trials comparing uncovered DSEMS and partially or fully covered DSEMS in patients with malignant GOO have reported comparable stent patency between the two types of stents.

Recently, the creation of a gastrojejunostomy under EUS (EUS-GJ) guidance using lumen-apposing stents has been described 12-16. The procedure was associated with a technical success rate of around 90% and clinical success of 85% to 100%. The procedure holds the potential to create a gastrojejunostomy without surgery. Furthermore, there is a low risk of tumor ingrowth and stent migration, thus improving the stent patency and reducing the need of re-intervention. However, there is limited data on how EPASS compares to endoscopic stenting. The aim of the current study is thus to compare prospective data on EPASS versus a historical group that received DSEMS.

DETAILED DESCRIPTION:
In recent years, DSEMSs have provided an attractive alternative to surgery for palliation of malignant gastric outlet obstruction. Several studies have assessed the clinical and technical success rates of DSEMS for malignant gastroduodenal obstruction. Technical success rates of 90% to 100% and clinical success of 80% to 95% was achieved.The procedure was associated with quicker recovery and reduced morbidities as compared to surgical gastrojejunostomies. However, the long-term patency of uncovered DSEMS is limited by the risk of tumor ingrowth that would lead to subsequent re-stenosis of the stents requiring re-intervention. Thus to palliate malignant gastric outlet obstruction, surgical gastrojejunostomy is preferred in patients that are fit for surgery with prolonged life expectancy whilst insertion of DSEMS is preferred in patients that are associated with high-risk for surgery and short life expectancy.

Recently, EUS-guided gastrojejunostomies have become possible. In the early description, a common technical problem exists in the series. The target duodenum or jejunum needed for creation of a GJ is collapsed and it is difficult to identify the target organ by EUS from the stomach. Furthermore, the insertion of the stent for creation of the anastomosis may be difficult with a collapsed bowel and this may result in catastrophic outcomes. To overcome this difficulty, our group has published the results of using the double balloon occluder that allows distension of the duodenum in conjunction with the AXIOS stent for creation of a GJ in 20 patients (Endoscopic ultrasonography-guided double-balloon-occluded gastrojejunostomy bypass - EPASS). The technical success rate was 90% (18/20). The median intubation time from the double-balloon tube intubation to stent placement was 25.5 min (range 10-39 min). Post-treatment gastric outlet obstruction scoring system (GOOSS) score improved in all 18 cases in which EPASS was successfully performed.

Thus, based on the above results, EUS-GJ may be associated with improved outcomes as compared with conventional procedures for management of malignant GOO. The aim of the current study is to compare the efficacies of EPASS in a prospective multicenter setting versus a historical cohort of uncovered DSEMS for patients suffering from unresectable malignant GOO.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients ≥ 18 years old
* Biopsy and/or cytology confirmed unresectable distal gastric or duodenal or pancreatico-biliary malignancies
* Suffering from gastric outlet obstruction with a gastric outlet obstruction score of ≤ 1 (appendix 1) 19 Performance status ECOG ≤3 (appendix 2)

Exclusion Criteria:

* Prior metallic stent placement
* Severe comorbidities precluding the endoscopic procedure (such as cardiopulmonary disease, sepsis, or a bleeding disorder)
* Life expectancy of less than 1 month
* History of gastric surgery
* Linitus plastic
* Multiple-level bowel obstruction confirmed on radiographic studies such as small bowel series or abdominal computed tomography
* Coagulation disorders
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2021-08-14 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
6 month re-intervention rate | 6 months
  percentage of patients requiring additional endoscopic intervention due to stent dysfunction

SECONDARY OUTCOMES:
technical success | 1 day
  successful placement of a stent across the site of obstruction, as confirmed by endoscopy or fluoroscopy
clinical success | 7 days
  improvement of at least 1 point in the GOOS within 3 days after stent insertion
adverse events rate | 30 days
  graded according to the lexicon of endoscopic adverse
mortality | 30 days
  Death within 30 day of the procedure
Post stenting gastric outlet obstruction scores | 7 days
  Degree of oral intake after stenting
the duration of stent patency | 6 months
  How long the stent remains patent
quality of life assessment scores | 6 months
  EORTC QLQ-C30

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Prince of Wales Hospital, Hong Kong, Hong Kong